CLINICAL TRIAL: NCT06915844
Title: Strengthening HPV Vaccination and Adolescent Health Research Program (SHARP) in Tanzania
Brief Title: Integrated HPV Vaccination and Adolescent Health in Tanzania
Acronym: SHARP-TZ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 30505
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Integrated Care; Adolescent; HPV

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive an adapted integrated adolescent health service package including HPV vaccination for 9-14 years, vision screening, nutritional services, comprehensive age-appropriate health education, appropriate screenings and referrals.
  Interventions: Behavioral: SHARP Tanzania
- Comparison (No Intervention): The comparison arm will receive routine adolescent health services including existing school-based integrated packages.

INTERVENTIONS:
Behavioral: SHARP Tanzania — Building on existing adolescent health services, including HPV+, this intervention adds desired services for adolescent health education, screening, counseling, and referrals. In addition, this intervention has strategic community engagement to identify out of school girls with limited access to existing integrated health services available in schools, community sensitization activities, and training for healthcare workers.
  Arms: Intervention

SUMMARY:
Background: Cervical cancer is a serious global public health problem, particularly in sub-Saharan Africa, where it is the leading cause of cancer in women, with around 70,722 new cases each year. Vaccination against human papillomavirus (HPV) prevents cervical cancer and is usually given to children around 9 to 15 years of age. HPV vaccination has been incorporated into many countries' Expanded Programs on Immunization, but often faces optimization and uptake challenges. SHARP is an implementation research initiative in Tanzania, Nigeria, and Côte d'Ivoire that is looking at the potential of combining HPV vaccination with with adolescent primary care/preventive health services - how this might work and its effect on the uptake of the HPV vaccine and other services.

Objective: To describe the feasibility, acceptability, effectiveness and sustainability of a locally-designed integrated adolescent health service package, including HPV vaccination in Tanzania. Specifically, this study aims to adapt an existing school based primary health care approaches, making service delivery not only more convenient but also more effective in addressing the specific needs of adolescents- focusing on out of school adolescents - in communities, and health facilities.

Methods: This is a quasi-experimental research study using a post intervention comparison approach to assess differences between an intervention group and a comparison group over time. It will use mixed methods drawing on quantitative surveys, qualitative interviews, service time motion assessment, and administrative data. The study will be conducted in two regions, each with an intervention and comparison district. The adapted adolescent integrated health intervention will be implemented in the intervention districts with routine service provision in comparison areas. Monthly administrative service coverage data and endline surveys will be conducted in up to 2880 households with 1400 parents/caregivers and 1600 adolescents will assess effectiveness by looking at changes in service uptake and coverage, as well in knowledge, attitudes, and practices towards HPV vaccination and integrated services. At endline, up to 68 in-depth interviews will be conducted with program managers, health officials, service providers, school authorities, community influencers and leaders, and adolescents and parents/caregivers will assess feasibility, acceptability and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents: Age: 9 to 15; Residence in the study regions; Parental or guardian permission is required; Provides assent and agrees to participate in the study.
* Parents/caregivers: Be the parent or legal guardian of an adolescent aged 9 to 15 years; Residence in the study regions; Provides informed consent and agrees to participate in the study.

Exclusion Criteria:

* People who have time constraints; participants who have medical conditions that make them unable to participate; those residing outside study health regions; those who do not provide consent/assent to participate.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number/proportion of adolescent girls vaccinated for HPV | Baseline (before intervention start) and at endline (after ~6 months intervention); monthly (program data)
  This is an effectiveness measure that captures the HPV coverage among adolescent girls residing in the study areas.
Number/proportion of adolescent girls intending to get HPV vaccine | Endline (after ~6 months intervention)
  This measure, captured through the survey, aggregates those who have received HPV vaccination in the past 6 months as well as those who express an intention to get vaccinated in the next 6 months.

SECONDARY OUTCOMES:
Number/proportion of participants with HPV knowledge | Endline (after ~6 months intervention)
  This measure will be captured through a survey by several knowledge related items, including a standardized composite measure.
Number/proportion of participants with positive attitudes towards integrated services | Endline (after ~6 months intervention)
  This outcome reflects several indicators related to attitudes related to accessing integrated adolescent health services, including HPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Sripad, PhD, MPH, Principal Investigator — Jhpiego
Locations (1):
- Muhimbili University of Health and Allied Sciences (MUHAS), Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No